CLINICAL TRIAL: NCT04769596
Title: Safety and Efficacy Study of the Neurent Medical NEUROMARK System in Subjects With Chronic Rhinitis A Double-blind, Sham Controlled Study
Brief Title: Safety and Efficacy Study of the Neurent Medical NEUROMARK™ System in Subjects With Chronic Rhinitis
Acronym: MERIDIEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurent Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLP-0005
Record Dates: First submitted 2021-02-15; First posted 2021-02-24 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Chronic Rhinitis
Keywords: Rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Sham Controlled Study
Who Masked: Participant
Masking Description: Subjects, site investigator, site personnel, and sponsor will be blinded to which study arm they are randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): Subject in this arm will undergo treatment with the NEUROMARK device.
  Interventions: Device: NEUROMARK™ System
- Sham (Sham Comparator): Subjects in this arm will undergo the procedure with a Sham device. At 3 months post treatment these subjects will cross over to Arm 1.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: NEUROMARK™ System — The NEUROMARK™ System is designed to deliver energy to the nasal cavity intended to interrupt nasal nerves aimed to reduce symptoms related to Chronic Rhinitis.
  Arms: Treatment
Device: Sham Device — A Sham device will be used in the nasal cavity
  Arms: Sham

SUMMARY:
A randomized, sham-controlled, double-blind study of the NEUROMARKTM system as a treatment for chronic rhinitis

DETAILED DESCRIPTION:
The MERIDIEN Study is a prospective, multi-center, double-blind, randomized (1:1), sham-controlled, cross-over study to evaluate the safety and efficacy of the NEUROMARK™ System in patients with Chronic Rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent, including authorization to release health information.
* Subject is 18 years of age or older at the time of consent.
* Subject has provided a negative pregnancy test (if Subject is a woman of childbearing potential (WOCBP).
* Subject WOCBP must be practicing and willing to continue an effective method of birth control during the course of the study.
* Subjects stated willingness to comply with all study procedures, post- treatment care and availability for the duration of the study follow up of 1 year.
* Subject tests negative for active COVID-19 at the start of study screening and continues to be free from COVID-19 symptoms until the time of enrollment/treatment.
* Subject understands and agrees to follow local COVID-19 restrictions (social distancing, face mask, etc.)

Exclusion Criteria:

* Subject has an allergy or intolerance to anaesthetic agent or other study-required materials.
* Subject is an active smoker or has been a smoker within the last 6 months (patient reported).
* Any physical condition that in the Investigator's opinion would prevent adequate study participation or pose increased risk to the study Subject.
* Subject is pregnant, nursing or plans to become pregnant during the study, or is a WOCBP, but is not willing to use an effective method of birth control.
* Patient is enrolled in an investigational drug or device study or has participated in such a study within the last 30 days prior to screening that in the opinion of the Investigator would interfere with the study results
* Patient presents with any condition or situation which, in the Investigator's opinion, puts the Subject at risk, could confound the study results, or may interfere significantly with the Subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Frequency of Serious Adverse Events (SAEs) directly attributable to the device | 1 month
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Annalise Sorensen, Study Director — Neurent Medical
Locations (8):
- United States (8):
  - Alabama Allergy, Birmingham, Alabama
  - Sacramento ENT, Roseville, California
  - Colorado ENT, Colorado Springs, Colorado
  - Tandem Clinical Research, Marrero, Louisiana
  - The Centers of Advanced ENT Care, Towson, Maryland
  - Specialty Physicians Associates, Bethlehem, Pennsylvania
  - Alamo ENT, San Antonio, Texas
  - Ear, Nose, Throat, & Allergy Associates, Puyallup, Washington

IPD SHARING:
Plan to Share IPD: No